CLINICAL TRIAL: NCT02708186
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Study of Nelotanserin Versus Placebo in Subjects With Dementia With Lewy Bodies (DLB) or Parkinson's Disease Dementia (PDD) Who Have REM Sleep Behavior Disorder (RBD)
Brief Title: Study Evaluating Nelotanserin for Treatment of REM Sleep Behavior Disorder in Subjects With Dementia (DLB or PDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Axovant Sciences Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sio Gene Therapies (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVT-102-2002
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Results first posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-04

CONDITIONS: Dementia With Lewy Bodies; REM Sleep Behavior Disorder; Parkinson's Disease Dementia
Keywords: Dementia with Lewy bodies; Lewy bodies; REM sleep behavior disorder; Parkinson's disease dementia
MeSH Terms: conditions — Lewy Body Disease; REM Sleep Behavior Disorder | interventions — nelotanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Nelotanserin (Experimental): Nelotanserin 80 mg
  Interventions: Drug: Nelotanserin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nelotanserin — once daily, oral, 20-mg tablets
  Arms: Nelotanserin
Drug: Placebo — once daily, oral, matching tablets
  Arms: Placebo

SUMMARY:
This study seeks to evaluate the safety and efficacy of Nelotanserin for the treatment of Rapid Eye Movement (REM) Sleep Behavior Disorder (RBD) in subjects with dementia with Lewy bodies (DLB) or Parkinson's disease dementia (PDD).

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, parallel-arm study in subjects with DLB or PDD who have RBD.

Subjects who meet the randomization criteria will be randomized 1:1 to receive Nelotanserin or placebo for 28 days during the double-blind period.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects at least 50 years of age, with a diagnosis of DLB or PDD and RBD based on Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) diagnostic criteria
* Presence of frequent REM sleep behavior episodes
* Mini Mental State Examination score ≥ 18

Exclusion Criteria:

* Subjects have a current diagnosis of significant psychotic disorders including, but not limited to, schizophrenia or bipolar disorder
* Subjects' RBD symptoms are secondary to or better accounted for by another medical condition, psychiatric disorder, or substance abuse
* Subjects with a current serious and/or unstable cardiovascular, respiratory, thyroid, gastrointestinal, renal, hematologic or other medical disorder

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilise Lombardo, MD, Study Director — Axovant Sciences, Inc., Clinical Research
Locations (23):
- United States (23):
  - US120, Birmingham, Alabama
  - US164, Phoenix, Arizona
  - US145, Sun City, Arizona
  - US143, Little Rock, Arkansas
  - US122, Englewood, Colorado
  - US180, Maitland, Florida
  - US154, Ocala, Florida
  - US113, Orlando, Florida
  - US152, Ormond Beach, Florida
  - US153, Tampa, Florida
  - US163, Atlanta, Georgia
  - US107, Indianapolis, Indiana
  - US132, Lenexa, Kansas
  - US129, Lincoln, Nebraska
  - US101, Chapel Hill, North Carolina
  - US159, New Bern, North Carolina
  - US147, Fargo, North Dakota
  - US111, Cincinnati, Ohio
  - US104, Cleveland, Ohio
  - US105, Columbus, Ohio
  - US173, Lincoln, Rhode Island
  - US128, Memphis, Tennessee
  - US131, San Antonio, Texas

REFERENCES:
- [Derived] Stefani A, Santamaria J, Iranzo A, Hackner H, Schenck CH, Hogl B. Nelotanserin as symptomatic treatment for rapid eye movement sleep behavior disorder: a double-blind randomized study using video analysis in patients with dementia with Lewy bodies or Parkinson's disease dementia. Sleep Med. 2021 May;81:180-187. doi: 10.1016/j.sleep.2021.02.038. Epub 2021 Feb 25. PMID 33714847

RESULTS

PARTICIPANT FLOW:
Groups:
- Nelotanserin: Nelotanserin 80 mg
  Nelotanserin: once daily, oral, 20-mg tablets. Dose will be titrated up to the 80 mg dose strength in a blinded fashion after an initial 5 days of treatment with 40 mg Nelotanserin.
Period: Overall Study
Arm/Group | Nelotanserin | Placebo
Started | 16 | 18
Completed | 14 | 16
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Population: The Safety population included subjects who took at least 1 dose of double-blind study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Nelotanserin | Placebo | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (6.37) | 72.2 (6.40) | 71.3 (6.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 5
  Male | 16 | 13 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 18 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in the Frequency of REM Sleep Behavior Disorders (RBD) From Baseline to the End of the Treatment Period (28 Days) Based on a Clinical Evaluator.
Description: The number of RBD (sum of simple/major and complex RBD events) per 10 minutes, based on video/audio assessment conducted at a sleep laboratory. Simple/major behaviors are jerks with higher movement amplitude, or intensity (e.g., whole body jerks, single limb jerk); Complex behaviors are Movements showing complexity of action and involving more muscle groups simultaneously or violent movements, and can be seen as the enactment of dream contents.
Time Frame: 28 days
Measure: Least Squares Mean (Standard Error); unit: Number of RBD per 10 min
Arm/Group | Nelotanserin | Placebo
Number analyzed (Participants) | 16 | 18
Number of RBD per 10 min | -1.47 (1.006) | -0.26 (1.027)

ADVERSE EVENTS:
Time Frame: 11 weeks
Arm/Group | Nelotanserin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 2/16 | 0/18
Other Adverse Events (participants affected / at risk) | 11/16 | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nelotanserin (N=16) | Placebo (N=18)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nelotanserin (N=16) | Placebo (N=18)
Anxiety (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT02708186/Prot_SAP_000.pdf